CLINICAL TRIAL: NCT02457169
Title: Addressing Systemic Health Disparities in Early ASD Identification and Treatment
Brief Title: Addressing Systemic Health Disparities in Early Identification and Treatment of Autism Spectrum Disorder (ASD): ABCD Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Tufts Medical Center (Other); Northeastern University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Abbey Eisenhower, Associate Professor, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMassBoston; 1R01MH104400-01 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-05-29 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent Engagement Intervention group (Experimental): This group of parents will receive the brief, 2-4 hour intervention which will utilize motivational interviewing principles to enhance parents' preschool engagement as their children transition from Early Intervention to preschool.
  Interventions: Behavioral: Parent Preschool Engagement intervention
- Attention Control (Other): Waitlist Control Group: This group will receive the brief, 2-4 hour intervention which will utilize motivational interviewing principles to enhance parents' preschool engagement as their children transition from Early Intervention to preschool after a 3 month delay.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Parent Preschool Engagement intervention — This 1-2 session intervention (2-4 hours total) will involve one-on-one session(s) for parents whose children (all of whom have received a diagnosis of ASD through our study) are turning 3 and therefore transitioning from the Early Intervention system to the public school special education system. The intervention will utilize motivational interviewing (MI) principles to equip parents with the skills, knowledge, and clarity of goals necessary to collaborate effectively with school special education staff and teachers, to advocate for their children's needs, and to be empowered to navigate the special education system.
  Arms: Parent Engagement Intervention group
Behavioral: Attention Control — The attention control condition is parallel in format (one-on-one between parent with interventionist) and intensity (1-2 sessions, or 2-4 hours total). It involves open-ended interviews with parents about their child's development and plans for school.
  Arms: Attention Control

SUMMARY:
The intervention under examination is designed to promote parents' school engagement following the transition from Early Intervention (EI) to preschool for parents of young children who were diagnosed with ASD through our screening and assessment protocol. The brief intervention employs principles of motivational interviewing to address not only the particular child characteristics and needs associated with ASD but also the unique, system-related challenges of navigating the special education system and advocating for appropriate services. Motivational interventions with parents are designed to elicit parents' specific, action-oriented goals for themselves and their children, enhancing motivation to pursue change, and addressing and resolving obstacles or sources of ambivalence.

By identifying and capitalizing on parents' strengths, empowering parents to develop specific goals, and improving parents' readiness to engage actively with their children's school, teacher, and educational team, we expect that this brief intervention will lead to higher levels of parental school involvement, higher special education engagement, and closer and more productive parent teacher relationships.

ELIGIBILITY:
Inclusion Criteria: Parents of children who participated in our screening and assessment study, whose children received diagnoses of autism through our assessment, AND

* whose children are turning 3 and transitioning out of Early Intervention services.

Exclusion Criteria: Children who are medically complex OR

* have a previous diagnosis of ASD outside of our study OR
* Don't have a parent/guardian who speak/understand sufficient English or Spanish to complete study materials OR
* Don't qualify for Early Intervention services

Ages: 14 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
parental school involvement | 3 months post-intervention
  parent report on the school involvement subscale of the Parent-Teacher Involvement Scale
parent-teacher relationship quality | 3 months post-intervention
  parent-report on the relationship subscale of the Parent-Teacher Involvement Scale
parent-special education engagement | 3 months post-intervention
  parent report on the Parent-Special Education Engagement Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Carter, PhD, Principal Investigator — University of Massachusetts, Boston

IPD SHARING:
Plan to Share IPD: No